CLINICAL TRIAL: NCT01520883
Title: Decisional Conflict and Needs Assessment in Shared Decision Making in Asthma Management
Brief Title: Evaluation of Decisional Conflict and Needs Assessment in Asthma Management
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); AllerGen NCE Inc. (Industry)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, Principal investigator, Laval University
Other Study IDs: CER 20646
Record Dates: First submitted 2011-10-04; First posted 2012-01-30 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DEcisional conflict

SUMMARY:
Many patients suffering from asthma are not compliant to their treatment and consequently, are not well controlled. Shared decision making intervention has shown an improvement in the outcome of patients with chronic disease. The aim of this study is to evaluate decisional conflict and to assess decisional needs of adults with asthma.

DETAILED DESCRIPTION:
Asthmatic patients will be recruited and asked to fill a decisional conflict scale.

Patients, asthma educators and physicians will also be recruited to fill a needs assessment questionnaire about decisions taken by asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* diagnosed asthma

Exclusion Criteria:

* received asthma education in the past 2 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with mild to moderate asthma controlled or slightly controlled
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measuring Decisional Conflict with a valid Decisional Conflict Scale | 6 month
  To measure the level of decisional conflict, subjects were asked to fill out a decisional conflict scale on asthma management which was developed by O'Connor adapted for our study. This questionnaire consisted of 16 questions. The answers used a Likert scale ranged from 1 - strongly agree to 5 - strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Quebec
Locations (1):
- Institut Universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada